CLINICAL TRIAL: NCT05039645
Title: A Pilot Study to Investigate the Use of Remote Thermovisual Monitoring in Patients With a Previous Diabetic Foot Ulcer, During the COVID-19 Pandemic.
Brief Title: Use of Remote Thermovisual Monitoring in Patients With a Previous Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bluedrop Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BMS CP001
Record Dates: First submitted 2021-06-04; First posted 2021-09-09 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The study is a single-arm, open-label, multicentre, pilot/feasibility study evaluating the adherence and usability of daily use of remote thermovisual monitoring alongside standard of care in patients with a previous DFU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Arm Study - All participants (Other): Study is open arm with no blinding or randomisation. Patients will receive standard care including frequent clinical visits, education, and preventative foot care/podiatry as required. Patients will also be given a DFS thermovisual scanner device. Patients will be instructed to use the DFS on a daily basis, at home, to record thermovisual data about the soles of their feet.
  Data collected from the DFS device will be transmitted to a remote, cloud-based server for daily review using the SRI software. If a temperature difference of >2.2°C between similar points on the left and right feet is identified for 2 consecutive scans, or visible signs of skin damage are observed, the site will be notified and sent a report containing the findings. Once notified the site will contact the patient by telephone and determine the best course of action based on standard practices (e.g. offloading, attending an appointment).
  Interventions: Behavioral: Patient specific, clinician determined Intervention

INTERVENTIONS:
Behavioral: Patient specific, clinician determined Intervention — Data collected from the DFS device will be transmitted to a remote, cloud-based server for daily review using the SRI software. If a temperature difference of >2.2°C between similar points on the left and right feet is identified for 2 consecutive scans, or visible signs of skin damage are observed, the site will be notified and sent a report containing the findings. Once notified the site will contact the patient by telephone and determine the best course of action based on standard practices (e.g. offloading, attending an appointment).

SUMMARY:
The goal of the clinical trial is to investigate adherence to, and effects of, the Bluedrop Monitoring System (BMS) in high-risk patients with at least one previous diabetic foot ulcer (DFU).

The BMS is a remote thermovisual monitoring system, which allows the condition of the soles of the feet to be remotely monitored for thermal and visual signs of inflammation, both of which may signal the onset of certain conditions, such as diabetic foot ulcers.

It is comprised of the Delta Foot Scanner (DFS) device and its accompanying Sentinel Review Interface (SRI) software.

The Covid-19 pandemic has driven the need for remote patient care where possible. Although this is challenging for people with foot ulcers, prevention is the key. Remote thermovisual monitoring might help reduce recurrent foot ulcers and therefore the number of necessary hospital visits which always puts the patient at increased risk of Covid infection.

DETAILED DESCRIPTION:
Despite the introduction of preventative foot care guidelines DFUs have a high re-ulceration rate. In the first 12 months following healing, 30-50% will develop a subsequent DFU and by year 5 this rate increases to 70%. Temperature monitoring has been proposed as a way to reduce this re-ulceration rate but has not been widely adopted.

Based on the existing evidence groups such as the International Working Group on the Diabetic Foot (IWGDF) have recommended temperature monitoring for the prevention of recurrent foot ulcers.

Despite these recommendations the technique has not been widely adopted. This is likely due to a number of factors, but NICE, in their guidance document for the prevention and management of foot ulcers (NG19) states:

"While temperature foot monitoring was found to be the only effective form of augmented self-examination, the intervention tool was felt to be quite difficult to use and required a strongly motivated population to actually perform consistently and fill out the required log books".

Bluedrop Medical have developed a product which leverages the existing evidence on temperature monitoring but builds it into a device which also includes the ability to take photographic images, is easy to use, and can integrate well with the healthcare system.

The goal of the clinical trial is to demonstrate that patients will use the device consistently over the course of the study. It will also be used to determine the clinician reported utility of thermovisual data to conduct a remote assessment or remote intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diabetes mellitus types 1 or 2
2. Aged 18 years or older
3. Have loss of protective sensation based on the presence of peripheral neuropathy (Vibration Perception Threshold (VPT) ≥ 25V on either foot)
4. Have a recent history of a DFU (i.e. an ulcer, defined as cutaneous erosion through the dermis on the foot) which was present for at least 2 weeks and has healed within 2-18 months before entry into the study
5. Ability to provide informed consent
6. Able to walk independently for 10m or more
7. The patient has foot care from a podiatrist or is willing to undergo foot care by a podiatrist
8. Access to a mobile phone so able to receive text notifications, or access to a landline to receive telephone call notifications.

Exclusion Criteria:

1. Active foot ulceration or open amputation sites
2. An ulcer that has deemed to have healed within the 2 months prior to entry into the study
3. Weight, when fully clothed, of greater than 150kg.
4. Active Charcot neuro-osteoarthropathy
5. Active foot infection
6. Any history of lower limb amputation
7. Significant Peripheral Arterial Disease (PAD) defined as history of revascularisation or absence of foot pulses
8. Concomitant severe physical or mental condition(s) that limit the ability to follow instructions for the study, based on the clinical judgment by the physician. This includes the inability to use DFS, without having a carer who can perform the temperature measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Patient Adherence | 3 months
  Patient adherence, tracked throughout duration of study, as measured through the number of device uses in each week, and the average number of device uses over the whole study.

SECONDARY OUTCOMES:
Clinic reported utility of thermovisual data for remote analysis and remote intervention - Number of scans in each Likert response category | 3 months
  On receipt of a report due to an identified issue the clinic will be asked to complete a brief survey to determine utility of thermovisual data to remotely assess and issue guidance to the patient. The survey will use a 5-point Likert scale to assess overall usefulness of the report for (1) remote analysis and (2) remote intervention. Responses will be scored from 1 (Strongly Disagree) to 5 (Strongly Agree), where larger scores indicate a more positive experience with the device.
  The number of scans in each Likert response category will be presented.
Clinic reported utility of thermovisual data for remote analysis and remote intervention - Percentage of scans in each Likert response category | 3 months
  On receipt of a report due to an identified issue the clinic will be asked to complete a brief survey to determine utility of thermovisual data to remotely assess and issue guidance to the patient. The survey will use a 5-point Likert scale to assess overall usefulness of the report for (1) remote analysis and (2) remote intervention. Responses will be scored from 1 (Strongly Disagree) to 5 (Strongly Agree), where larger scores indicate a more positive experience with the device.
  The percentage of scans in each Likert response category will be presented.
Level of agreement between in-person visual assessment and remote assessment. | 3 months
  When the patient reports for a scheduled or unscheduled visit the clinic will carry out an in-person visual assessment of the feet. Visible signs of skin damage on the plantar surface of the feet will be recorded. In addition to this, at the end of the study, a blinded clinician will retrospectively review the 4 thermovisual scans taken prior to the schedule or unscheduled visit and record any signs of skin damage. The level of agreement between the in-person visual assessment and the remote assessment using the scans will then be determined.Identified skin issues in both the in-person and remote assessments will be categorized and grouped together using headings such as DFU, callus, discoloration, deformation. The location of the issue will also be recorded (e.g. plantar surface, interdigit, etc).
  The degree of agreement between the dichotomous scores from in-person visual assessment and the remote scan assessment will be determined using Cohen's kappa (κ).
Patient reported device usability | 3 months
  Patient reported device convenience, ease of use, usefulness of text reminders, impact on attitude towards care and overall satisfaction will be assessed via a survey during, and at the end, of the study.
DFU Incidence rates and severities | 3 months
  DFU severity will be assessed using the Texas wound classification system and the SINBAD scale. The relative depth of the ulcer, presence of infection or ischaemia or both will be used to categorise the wound grade and stage. The SINBAD Classification System assigns a SINBAD score from 0 to 6 to each ulcer based on a set of criteria, and larger scores indicate more severe ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Boulton, PhD, Principal Investigator — Prof. of Medicine, University of Manchester & Consultant Physician, Manchester Royal Infirmary; Caroline McIntosh, PhD, Principal Investigator — Podiatric Medicine School of Health Sciences Áras Moyola, NUI Galway
Locations (2):
- Merlin Park University Hospital, Galway, Ireland
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Armstrong DG, Athanasiou KA, Agrawal CM. Home monitoring of foot skin temperatures to prevent ulceration. Diabetes Care. 2004 Nov;27(11):2642-7. doi: 10.2337/diacare.27.11.2642. PMID 15504999
- [Background] Lavery LA, Higgins KR, Lanctot DR, Constantinides GP, Zamorano RG, Athanasiou KA, Armstrong DG, Agrawal CM. Preventing diabetic foot ulcer recurrence in high-risk patients: use of temperature monitoring as a self-assessment tool. Diabetes Care. 2007 Jan;30(1):14-20. doi: 10.2337/dc06-1600. PMID 17192326
- [Background] Armstrong DG, Holtz-Neiderer K, Wendel C, Mohler MJ, Kimbriel HR, Lavery LA. Skin temperature monitoring reduces the risk for diabetic foot ulceration in high-risk patients. Am J Med. 2007 Dec;120(12):1042-6. doi: 10.1016/j.amjmed.2007.06.028. PMID 18060924
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Abbott CA, Carrington AL, Ashe H, Bath S, Every LC, Griffiths J, Hann AW, Hussein A, Jackson N, Johnson KE, Ryder CH, Torkington R, Van Ross ER, Whalley AM, Widdows P, Williamson S, Boulton AJ; North-West Diabetes Foot Care Study. The North-West Diabetes Foot Care Study: incidence of, and risk factors for, new diabetic foot ulceration in a community-based patient cohort. Diabet Med. 2002 May;19(5):377-84. doi: 10.1046/j.1464-5491.2002.00698.x. PMID 12027925
- [Background] Boulton AJ, Kirsner RS, Vileikyte L. Clinical practice. Neuropathic diabetic foot ulcers. N Engl J Med. 2004 Jul 1;351(1):48-55. doi: 10.1056/NEJMcp032966. No abstract available. PMID 15229307
- [Background] Kerr M, Barron E, Chadwick P, Evans T, Kong WM, Rayman G, Sutton-Smith M, Todd G, Young B, Jeffcoate WJ. The cost of diabetic foot ulcers and amputations to the National Health Service in England. Diabet Med. 2019 Aug;36(8):995-1002. doi: 10.1111/dme.13973. Epub 2019 Jun 5. PMID 31004370
- [Background] Bus SA, van Netten JJ, Lavery LA, Monteiro-Soares M, Rasmussen A, Jubiz Y, Price PE; International Working Group on the Diabetic Foot. IWGDF guidance on the prevention of foot ulcers in at-risk patients with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:16-24. doi: 10.1002/dmrr.2696. No abstract available. PMID 26334001
- [Background] Bus SA, van Netten JJ. A shift in priority in diabetic foot care and research: 75% of foot ulcers are preventable. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:195-200. doi: 10.1002/dmrr.2738. PMID 26452160
- [Background] Jeffcoate WJ, Vileikyte L, Boyko EJ, Armstrong DG, Boulton AJM. Current Challenges and Opportunities in the Prevention and Management of Diabetic Foot Ulcers. Diabetes Care. 2018 Apr;41(4):645-652. doi: 10.2337/dc17-1836. PMID 29559450
- [Background] Yap MH, Chatwin KE, Ng CC, Abbott CA, Bowling FL, Rajbhandari S, Boulton AJM, Reeves ND. A New Mobile Application for Standardizing Diabetic Foot Images. J Diabetes Sci Technol. 2018 Jan;12(1):169-173. doi: 10.1177/1932296817713761. Epub 2017 Jun 21. PMID 28637356